CLINICAL TRIAL: NCT01859533
Title: Positive End Expiratory Pressure With A T-piece Resuscitator (Neopuff) For Near-Term and Term Infants With Respiratory Distress: A Randomized, Controlled Trial
Brief Title: Positive End Expiratory Pressure With A T-piece Resuscitator For Near-Term and Term Infants With Respiratory Distress
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Ali El-Farrash, Lecturer of Pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ain Shams Uni
Record Dates: First submitted 2013-05-16; First posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Transient Tachypnea of the Newborn
MeSH Terms: conditions — Transient Tachypnea of the Newborn

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neopuff group (Experimental): includes 34 newborns showing signs of TTN who received CPAP (5 cm of H2O) via T- piece (Neopuff; Fisher and Paykel Healthcare, Auckland, New Zealand).
  Interventions: Device: Neopuff
- Control group (No Intervention): includes 30 newborns who will receive nasal prong oxygen treatment; standard care according to Siva Subramanian et al. (2010).

INTERVENTIONS:
Device: Neopuff — * Group I neonates (Experimental group) includes 30 newborns showing signs of TTN who will receive administration of CPAP (5 cm of H2O) via T- piece (Neopuff; Fisher and Paykel Healthcare, Auckland, New Zealand).
  * Group II neonates (Control group) includes 30 newborns who will receive nasal prong oxygen treatment; standard care according to Siva Subramanian et al. (2010).
  Other Names: Early CPAP
  Arms: Neopuff group

SUMMARY:
Evaluating the effect of early application of Continuous positive airway pressure (CPAP) via Neopuff in cases of transient tachypnea of the newborn(TTN) and its role in decreasing the duration and complication of TTN.

DETAILED DESCRIPTION:
The aim of the study is to determine whether positive end expiratory pressure therapy (PEEP) administered early via a T piece based infant resuscitator (Neopuff) would safely reduce the incidence of TTN and the need for neonatal intensive care unit (NICU) admission of near term and term infants with respiratory distress.

ELIGIBILITY:
Inclusion Criteria:

* Near term infants (36-37 weeks gestational age) and Full term infants (38-41 weeks gestational age).
* Presence of signs of respiratory distress (Tachypnea, intercostal and subcostal retractions, nasal flaring and grunting) evident shortly after birth.
* Cesarean section (CS) was defined as elective when surgery was performed before the onset of labor, with all other cases defined as secondary CS.

Exclusion Criteria:

* Presence of any of the risk factors for neonatal sepsis such as Prolonged Rupture of Membranes for ≥48 hours (PROM), maternal fever, maternal chorioamnionitis or positive maternal GBS colonization.
* Presence of any other cause of respiratory distress, eg.

  * congenital malformations affecting the cardiorespiratory system ,
  * chromosomal aberrations,
  * depression at birth (Apgar score at 5 minutes of < 7 or umbilical artery pH of < 7.10),
  * fetal hydrops,
  * persistent pulmonary hypertension,
  * and meconium aspiration syndrome.

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2011-11; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Need for admissions to NICU secondary to TTN | 24 hours

SECONDARY OUTCOMES:
Levels of plasma brain natriuretic peptide and clinical outcome [Time Frame: 24 hours]. | 24 hours
Duration of tachypnea. | until discharge
Duration and type of oxygen therapy. | ntil discharge
Antibiotic treatment. | until discharge
Incidence of pulmonary air leaks | ntil discharge
Length of hospital (NICU) stay | until discharge
Death | until discharge

CONTACTS AND LOCATIONS:
Overall Officials: Rania A. El-Farrash, MD, PhD, Principal Investigator — Associate Professor of Pediatrics, Department of Pediatrics, Ain Shams University, Cairo, Egypt; Amani O. Mahmoud, MD, Study Chair — Professor of Pediatrics, Department of Pediatrics, Ain Shams University, Cairo, Egypt; Enas H. Abdul-Hady, M.B.B.Ch, Principal Investigator — Ministry of Health